CLINICAL TRIAL: NCT01180049
Title: A RANDOMIZED PHASE 4 STUDY COMPARING 2 INTRAVENOUS TEMSIROLIMUS (TEMSR) REGIMENS IN SUBJECTS WITH RELAPSED, REFRACTORY MANTLE CELL LYMPHOMA
Brief Title: Comparison Of 2 Doses Of Temsirolimus (Torisel) In Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-4438; B1771007 (Other: Alias Study Number); 2009-015498-11 (EudraCT Number)
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; temsirolimus
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- temsirolimus (Torisel) 175mg weekly x 3, then 75mg weekly (Active Comparator)
  Interventions: Drug: temsirolimus
- temsirolimus (Torisel) 75mg weekly (Active Comparator)
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus — 175mg IV once a week for first 3 weeks, followed by 75mg IV once a week until disease progression, provided that patient is tolerating treatment and getting clinical benefit
  Other Names: Torisel
  Arms: temsirolimus (Torisel) 175mg weekly x 3, then 75mg weekly
Drug: temsirolimus — 75mg IV once a week until until disease progression, provided that patient is tolerating treatment and getting clinical benefit
  Other Names: Torisel
  Arms: temsirolimus (Torisel) 75mg weekly

SUMMARY:
This study will compare the effectiveness and safety of two different doses of temsirolimus (Torisel).

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed mantle cell lymphoma diagnosis.
* Have measurable disease.
* Have received at least 2 prior treatment, which may include stem cell transplant.
* Have adequate organ and bone marrow function.
* There are other criteria--please discuss with your doctor.

Exclusion Criteria:

* Had any prior treatment with temsirolimus or mTOR inhibitor.
* Had allogeneic stem cell transplant within last 6 months and on immunosuppressive therapy.
* Has active or untreated brain or central nervous system metastases.
* There are other criteria--please discuss with your doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (6):
  - Mercy Research Institute, Miami, Florida
  - Veterans Affairs New Jersey Healthcare System-Hematology/Oncology Section (111), East Orange, New Jersey
  - Mercy Clinic Oklahoma Communities dba Mercy Clinic Oncology/Hematology-McAuley, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City-Oncology Infusion, Oklahoma City, Oklahoma
  - Amy Shen, RPh, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
- Australia (5):
  - St George Hospital, Kogarah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Czechia (3):
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Czech Republic
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- CHU de Nancy, Vandœuvre-lès-Nancy, France
- Germany (2):
  - Klinik fuer Onkologie und Haematologie, Medizinische Klinik IV, Aachen
  - Klinikum Johannes-Gutenberg -Universitaet, III. Medizinische Klinik und Poliklinik, Mainz
- Italy (3):
  - Presidio Ferrarotto - A.O.U. - PoliclinicoVittorio Emanuele, Catania
  - Dipartimento di Medicina Diagnostica, Clinica e di Sanità Pubblica, Modena
  - Struttura Complessa di Ematologia, Dipartimento di Oncologia ed Ematologia-, Torino
- Malopolskie Centrum Medyczne S.C., Krakow, Poland
- Romania (3):
  - Institutul Clinic Fundeni Bucuresti, Sectia II Hematologie, Bucharest
  - Spitalul Clinic Coltea, Clinica de Hematologie, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Clinica de Hematologie, Bucharest
- Russia (3):
  - Republican Clinical Oncology Dispensary of the Ministry of Healthcare of Tatarstan Republic, Kazan'
  - GBOU VPO "First Saint-Petersburg State Medical University n.a. I.P.Pavlov", Saint Petersburg
  - Institute of Pediatric Hematology and Transplantology R.M.Gorbacheva, Saint Petersburg
- Serbia (2):
  - Clinical Centre of Serbia,Clinic for Hematology, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- South Korea (2):
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-4438&StudyName=Comparison%20Of%202%20Doses%20Of%20Temsirolimus%20%28Torisel%29%20In%20Patients%20With%20Mantle%20Cell%20Lymphoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers from 10 Mar 2011 to 28 Jun 2018.
Groups:
- TEMSR 175/75 mg: Participants had received desipramine 50 milligrams (mg) one week prior to the first dose of temsirolimus (TEMSR). An additional desipramine 50 mg was administered again approximately 30 min prior to every first dose of TEMSR on Day 1. Participants then received 175 mg intravenously (IV) once weekly for the first 3 weeks and followed by 75 mg once weekly thereafter.
- TEMSR 75 mg: Participants had received desipramine 50 mg one week prior to the first dose of TEMSR. An additional desipramine 50 mg was administered again approximately 30 min prior to every first dose of TEMSR on Day 1. Participants then received TEMSR 75 mg IV once weekly.
Period: Overall Study
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Started | 53 | 48
Completed | 0 | 0
Not Completed | 53 | 48
Not completed — Other | 9 | 7
Not completed — Lost to Follow-up | 8 | 6
Not completed — Death | 36 | 35

BASELINE CHARACTERISTICS:
Population: The analysis was done on Intent-to-Treat (ITT) Population which included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug dose from that to which they were randomized.
Groups:
- TEMSR 175/75 mg: Participants had received desipramine 50 mg one week prior to the first dose of temsirolimus (TEMSR). An additional desipramine 50 mg was administered again approximately 30 min prior to every first dose of TEMSR on Day 1. Participants then received 175 mg IV once weekly for the first 3 weeks and followed by 75 mg once weekly thereafter.
- Total: Total of all reporting groups
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg | Total
Number analyzed (Participants) | 53 | 48 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (9.11) | 66.3 (8.36) | 66.8 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Independently Assessed Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to first documentation of disease progression by the independent assessor or to death due to any cause, whichever occurred first.
  PFS = (earliest date of progression or death due to any cause- randomization date+1)/30.4.
  PFS assessment was done using EMA guidelines for sensitivity analysis censoring.
  Participants who were alive and progression-free at the time of analysis were censored on the date of last assessment; participants without adequate baseline assessment or without post-baseline assessments were censored on the randomization date; participants who died or progressed after 2 or more missed visits were censored on the date of last tumor assessment prior to the missing visit; and participants who started new anti-cancer therapy prior to death or progression were censored on the date of last tumor assessment prior to the start of anti-tumor treatment.
Time Frame: From randomization date to the date of first documentation of progression or death (average follow up done for 15 months)
Population: The analysis was done on ITT population which included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug dose from that to which they were randomized.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 47 | 43
Months | 4.3 [3.3 to 6.4] | 4.5 [2.7 to 4.9]
Statistical Analysis 1: Comparison: TEMSR 175/75 mg vs TEMSR 75 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 0.731, 80% CI 2-sided [0.520 to 1.027]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From randomization date until death due to any cause (average follow up done for 56.1 months)
Population: Analysis was done on ITT population. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 53 | 48
Months | 10.9 [7.0 to 19.7] | 11.2 [6.6 to 18.1]
Statistical Analysis 1: Comparison: TEMSR 175/75 mg vs TEMSR 75 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 0.778, 80% CI 2-sided [0.568 to 1.064]

3. Secondary Outcome: Independent Assessment - Objective Response Rate (ORR = CR + PR)
Description: ORR is defined as the percentage of participants with confirmed CR or PR according to the Cheson Criteria relative to all randomized Participants. Tumor responses were determined using information from objective measurements from computed tomography information including B-symptom evaluation, physical examination, ECOG performance status, assessment of liver and spleen, laboratory assessments such as bone marrow biopsies and/or aspirates, biochemical markers of disease activity and hematology results.
  Participants who did not have on-study radiographic tumor re-evaluation or who died, progressed or dropped out for any reason prior to reaching a CR or PR were counted as non-responders in the (CT) scans, as well as clinical assessment of ORR.
Time Frame: From randomization date until end of treatment (average follow up done for 15 months)
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 47 | 43
Percentage of participants | 27.7 [19.1 to 37.7] | 20.9 [13.0 to 31.0]
Statistical Analysis 1: Comparison: TEMSR 175/75 mg vs TEMSR 75 mg; Independent assessment- Difference (%) TEMSR 175/75 mg - TEMSR 75 mg (80% CI); Test type: Superiority or Other; Difference in arms = 6.7, 80% CI 2-sided [-6.9 to 20.3]

4. Secondary Outcome: Investigator's Assessment ORR (ORR = CR + PR)
Description: as for outcome 3
Time Frame: From randomization date until end of treatment (average follow up done for 15 months)
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 47 | 43
Percentage of participants | 31.9 [22.9 to 42.2] | 18.6 [11.1 to 28.5]
Statistical Analysis 1: Comparison: TEMSR 175/75 mg vs TEMSR 75 mg; Investigator's assessment- Difference (%)TEMSR 175/75 mg - TEMSR 75 mg (80% CI); Test type: Superiority or Other; Difference between arms = 13.3, 80% CI 2-sided [-0.4 to 26.7]

5. Secondary Outcome: Investigator Assessed PFS
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 47 | 43
Months | 4.7 [2.7 to 8.3] | 3.9 [2.8 to 4.7]
Statistical Analysis 1: Comparison: TEMSR 175/75 mg vs TEMSR 75 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 0.646, 80% CI 2-sided [0.453 to 0.922]

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Infection- Related Adverse Events (AEs) With Grade 2 or Higher as Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Treatment emergent adverse event=as an event that emerged during treatment period that was absent before treatment, or worsened during treatment period relative to pretreatment state. Treatment-emergent infection-related AEs included events: pneumonia, bronchitis, infection, herpes simplex, oral candidiasis and sepsis. Grading by NCI CTCAE Version 3.0.: Grade 1= mild; Grade 2= moderate; Grade 3= severe; Grade 4= life-threatening; urgent intervention indicated; Grade 5= death.
Time Frame: From screening up to a maximum of 57.1 months
Population: Analysis was done on safety population which included any participant who received at least 1 dose of TEMSR was included in the evaluation for safety.
Measure: Number; unit: Percentage of participants
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 53 | 47
Percentage of participants
  Pneumonia | 17.0 | 21.3
  Bronchitis | 7.5 | 2.1
  Infection | 5.7 | 2.1
  Herpes simplex | 3.8 | 2.1
  Oral candidiasis | 3.8 | 0
  Cellulitis | 1.9 | 0
  Sepsis | 0 | 2.1

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Bleeding-Related AEs With Grade 2 or Higher as Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Treatment emergent adverse event=as an event that emerged during treatment period that was absent before treatment, or worsened during treatment period relative to pretreatment state. Treatment-emergent bleeding related AEs included events: epistaxis and ecchymosis. AE were assessed according to maximum severity grading based on NCI CTCAE Version 4.03.Grade 1=mild; Grade 2=moderate; within normal limits. Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening or disabling; urgent intervention indicated; Grade 5=death.
Time Frame: From screening up to a maximum of 57.1 months
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 53 | 47
Percentage of participants
  Epistaxis | 13.2 | 2.1
  Ecchymosis | 1.9 | 0

8. Secondary Outcome: Quantify the Potential Effect of TEMSR on AUC and Cmax
Description: Potential TEMSR effects were investigated by calculating the ratio of AUCs with and without concomitant TEMSR from the model-estimated effect of TEMSR on apparent clearance (CL/F) values and using individual ratios of observed Cmax values with and without concomitant temsirolimus, for both parent and metabolite. The AUC mean ratio was calculated as 1 / mean shift on apparent clearance from TEMSR, and the 90% CI of the AUC ratios was calculated as 1 / 90% CI of the shift on apparent clearance from TEMSR.
  AUC: Area under plasma concentration-time curve from time zero to infinity Cmax: Characterization of maximum observed plasma concentration
Time Frame: From one week predose (Day -7, -4hr, -8hr, -48hr) upto 2 weeks post dose (4hr, 8hr, 48hr and Day 8)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Ratio
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Number analyzed (Participants) | 47 | 43
Ratio
  AUC | 1.00 [0.965 to 1.11] | 0.980 [0.870 to 1.12]
  Cmax | 0.828 [0.758 to 0.898] | 0.779 [0.7005 to 0.857]

ADVERSE EVENTS:
Time Frame: From screening up to a maximum of 57.1 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis was done on safety population which included any participant who received at least 1 dose of TEMSR.
Arm/Group | TEMSR 175/75 mg | TEMSR 75 mg
Serious Adverse Events (participants affected / at risk) | 35/53 | 34/47
Other Adverse Events (participants affected / at risk) | 51/53 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEMSR 175/75 mg (N=53) | TEMSR 75 mg (N=47)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 10 | 9
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 1
Bronchitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Fungal infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Listeria sepsis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 9
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Viral skin infection (Infections and infestations) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Haemoglobin (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cataract (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Human rhinovirus test positive (Investigations) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEMSR 175/75 mg (N=53) | TEMSR 75 mg (N=47)
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Leukopenia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 18 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 37 | 28
Tachycardia (Cardiac disorders) | 0 | 4
Dry eye (Eye disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 19 | 14
Mouth ulceration (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 9
Stomatitis (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 7 | 7
Chest discomfort (General disorders) | 1 | 4
Fatigue (General disorders) | 11 | 13
Decreased appetite (Metabolism and nutrition disorders) | 6 | 8
Oedema peripheral (General disorders) | 9 | 8
Pyrexia (General disorders) | 13 | 11
Bronchitis (Infections and infestations) | 4 | 1
Herpes simplex (Infections and infestations) | 4 | 2
Infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 3 | 4
Rhinitis (Infections and infestations) | 4 | 1
Skin infection (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 10 | 10
Urinary tract infection (Infections and infestations) | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Blood pressure increased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 6 | 2
Weight decreased (Investigations) | 6 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 5 | 3
Initial insomnia (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 5 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 10 | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 3 | 0
Mucosal inflammation (General disorders) | 3 | 5
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 4
Oral candidiasis (Infections and infestations) | 3 | 2
Blood cholesterol increased (Investigations) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
Overall Survival was not collected for the intended duration as planned initially, no long term follow up was conducted according to amendment in protocol. Hence overall survival results were limited

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.